CLINICAL TRIAL: NCT01792401
Title: Probiotics in Enteral Feeding in Critically Ill Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Ausama A Malik, Surgeon/Clinical Specialist, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEFCIP
Record Dates: First submitted 2013-02-08; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Critical Illness; Dietary Modification; Probiotics; Gut Failure; Treatment Outcomes
Keywords: Critical illness; Dietary supplements; Gastrointestinal tract/physio-pathology
MeSH Terms: conditions — Critical Illness | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Patients on enteral feeding in intensive care units are administered a placebo
  Interventions: Drug: Placebo
- Probiotics (Active Comparator): Patients on enteral feeding in intensive care unit are given a probiotic
  Interventions: Drug: Probiotics

INTERVENTIONS:
Drug: Probiotics
  Arms: Probiotics
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of probiotics in enteral nutrition on improving gut function, inflammatory markers and clinical outcomes in critically ill patients admitted to the intensive care unit.

DETAILED DESCRIPTION:
Gut failure in critically ill patients is common. Enteral feeding is one of the preferred routes for nutrition support to maintain gut function. However, enteral nutrition is not without complications such as alterations in gut transit time and gut eco-culture. Enteral nutrition supplemented with a probiotic offers a possible solution to modulating this ecosystem. Objectives: The primary aim of this study was to investigate the effect of probiotics in enteral feeding on improving the gut function, inflammatory markers and clinical outcomes in critically ill patients. Subjects and Methods: Forty-nine patients that were admitted to the intensive care unit in University Malaya Medical Center requiring enteral feeding were randomized to receive either probiotics or a placebo. Patients remained in the intensive care unit for more than 7 days and were examined prior to the start of enteral feeding and on day 8. Return of gut function was assessed by the time needed to achieve caloric requirement. Inflammatory markers including the White Cell Count and C-reactive protein levels were tested on day 1 and day 8. Clinical outcome was assessed by number of days of ventilation and total days in intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to intensive care unit
* Expected stay of more than 48 hours
* On enteral feeding
* Consent obtained from patient/relative

Exclusion Criteria:

* Patients on immuno-suppressive drugs
* Patients with hematological diseases
* Pregnant females
* Do not consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Improve the time to return of gut function in patient on enteral feeding in intensive care unit | Time required to achieve maximum enteral feeding with a minimum of 48 hours
  Probiotic/placebo administered once enteral feeding is started, and the hours needed to achieve maximum feeding is calculated in hours

SECONDARY OUTCOMES:
Inflammatory markers | 7-14 days
  Measure of inflammatory markers are obtained from patients at the start and at the end of probiotic/placebo administrations.

OTHER OUTCOMES:
Clinical Outcome | Patients will be followed up throughtout their duration of intensive care stay, or a minimum of 1-14 days
  Number of days in intensive care and number of ventilation days are calculated at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ausama A Malik, MS,MBBS(Mal), Principal Investigator — University Malaya Medical Center; Kin Fah Chin, FRCS (Glasg), Study Chair — University of Malaya; Vineya Rai Hakumat Rai, M. Anes,MBBS, Study Chair — University of Malaya; Chee Loong Yeap, MS,MBBS(Mal), Study Chair — University of Malaya; Peng Choong Lau, MS,MBBS(Mal), Study Chair — University of Malaya; Eng Hong Pok, MS,MBBS(Mal), Study Chair — University of Malaya; Gowri Rajandram, Phd(Aust), Study Chair — University of Malaya
Locations (1):
- University Malaya Medical Center, Kuala Lumpur, Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] Malik AA, Rajandram R, Tah PC, Hakumat-Rai VR, Chin KF. Microbial cell preparation in enteral feeding in critically ill patients: A randomized, double-blind, placebo-controlled clinical trial. J Crit Care. 2016 Apr;32:182-8. doi: 10.1016/j.jcrc.2015.12.008. Epub 2015 Dec 15. PMID 26777745